CLINICAL TRIAL: NCT06401850
Title: Training Given to Women With Polycystic Ovary Syndrome Effect on Quality of Life: A Randomized Controlled Study
Brief Title: Polycystic Ovary Syndrome and Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: pcos
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life
Keywords: Polycystic Ovary Syndrome; Quality of Life; Education
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): Training for women with Polycystic Ovary Syndrome (POS) can play an important role in improving quality of life and managing symptoms. These trainings may cover topics such as healthy lifestyle choices, nutritional habits, exercise, stress management and strategies to support hormone balance. Acquiring these knowledge and skills can help women cope with POS, promote psychosocial recovery, and improve their overall quality of life.
  Interventions: Other: Education Group
- Control Group (Experimental): Since there was no training given to the control group, its effect on the participants' quality of life could not be evaluated. However, considering the potential of regularly provided training for women with polycystic ovary syndrome to improve quality of life, it may be important to provide similar training to the control group and compare the results. In this way, the effectiveness of training can be understood more clearly and the relationship between POS and quality of life can be evaluated more comprehensively.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Education Group — The intervention provided to the training group focuses on improving skills to cope with polycystic ovary syndrome. This intervention includes topics such as encouraging healthy lifestyle habits, raising awareness about nutrition and exercise, teaching stress management techniques, and offering strategies to support hormonal balance. It provides participants with the tools they need to understand and manage symptoms that impact their lives. It also provides a supportive environment, encouraging participants to share their experiences with each other and receive support. This intervention aims to improve individuals' overall quality of life while strengthening their ability to manage their own health and well-being.
  Arms: Education Group
Other: Control Group — No intervention was made to the control group. This group did not receive additional training or support to cope with polycystic ovary syndrome. In this way, the effects of the control group on lifestyle, symptom management and overall quality of life were evaluated in comparison with the training group. This approach focuses on determining the direct effects of the intervention, while allowing to observe the natural course of the control group, and the results help to provide a clear assessment of the effectiveness of the intervention.
  Arms: Control Group

SUMMARY:
Aim: This research is being designed to determine the effect of Polycystic Ovary Syndrome (PCOS) education given to women on their quality of life. In this context, the aim of the project is; The aim is to determine the impact of the education given to women with PCOS on the quality of life of the training given to women with the disease, such as psychosocial and emotional status, fertility, sexual function, obesity and menstrual irregularity, and hair growth.

Method: Within the scope of this research, quantitative research method is used as the research method. In addition, it is planned as a randomized controlled quasi-experimental, which is one of the quantitative research methods. In calculating the sample size, type 1 error, research power and effect size parameters are determined before the research begins. Studies generally need to have at least 80% power. In order to find a significant difference, it is calculated that there should be at least 30 students in each group at 80% power and 95% confidence level. Considering the possible risks, it is planned to include 70 women in total in 2 groups (study and control), with 35 women in each group. All individuals who want to respond to the survey are included in the sample. The process of finding a subject continues until the desired size is reached. In addition, during the data collection process, participants were asked; They are asked whether they are diagnosed with PCOS and those who answer "yes" are included in the sample. Within the scope of the research, the voluntariness of the participants is essential and both written and verbal consents are obtained from each participant through an informed consent form. "Personal Information Form" and "Polycystic Ovary Syndrome Quality of Life-50 Scale" created by the researchers were used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

Individuals who are over 18 years of age, open to communication, diagnosed with PCOS, have no mental problems that require treatment, have no physical, mental or five sense disabilities, speak Turkish and can read and write, and volunteer to participate in the study.

Exclusion Criteria:

Individuals who are under 18 years old, not open to communication, diagnosed with PCOS, require treatment for significant mental health issues, have physical, mental, or sensory impairments, cannot speak or read and write Turkish, and are not willing to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because PCOS occurs in women.
Enrollment: 70 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life grade | before and 3 months after education
  To evaluate the impact on the quality of life of entrepreneurs. PCOS-50 standard questionnaires, one of the widely used scales, can be used to determine the quality of life of women with polycystic ovary syndrome. PCOS-50 allows participants to self-assess themselves in a variety of areas, including physical health, mental health, social functioning, pain, and general well-being. This scale is widely accepted for objectively assessing the impact of intervention on managing polycystic ovary syndrome symptoms and improving quality of life. This outcome measure provides a key criterion for evaluating the effectiveness of the intervention and enables outcomes to be measured in a scientifically valid and reliable manner.

CONTACTS AND LOCATIONS:
Overall Officials: Rüveyda Ölmez Yalazı, PhDc, Principal Investigator — Marmara University; Nurdan Demirci, Prof, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No